CLINICAL TRIAL: NCT03358615
Title: Robson Classification of Indications of Cesarean Section at a University Hospital in Egypt
Brief Title: Robson Classification of Indications of Cesarean Section at MUH
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hanan Nabil, Assistant Professor, Mansoura University
Other Study IDs: Robsen classification
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Indication of Cesarean Section
Keywords: robson classification; Egypt
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cesarean section — assessment of the indications of cesarean section according to Robson criteria

SUMMARY:
Robson classification of Cesarean section rates and indications allows evaluation and comparison of the contributors to the Cesarean section rate and their impact. It also allows comparison between institutions, regions, and countries that adopt this classification Robson's system classifies all deliveries into one of ten groups on the basis of five parameters: obstetric history (parity and previous cesarean section), onset of labor (spontaneous, induced, or cesarean section before onset of labor), fetal presentation or lie (cephalic, breech, or transverse), number of neonates, and gestational age (preterm or term; panel This study evaluates C.S rates and indications according to Robson classification in a University Hospital in a year (2016) to compare with international standards

ELIGIBILITY:
Inclusion Criteria:

* all cases who underwent CS at Mansoura University Hospital inpatients and emergency cases

Exclusion Criteria:

* non

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective study of an obstetric ,for booked (inpatient), non-booked (emergency) cases.
  Full data sheet- from for the case (history, examination, diagnosis, pregnancy duration ,labor onset: spontaneous or induced , and previous pregnancy C.S or not
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of C.S rates and indications according to Robson classification | one year
  comparison of the results with the international standards

CONTACTS AND LOCATIONS:
Locations (1):
- mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No